CLINICAL TRIAL: NCT00190905
Title: Study of Duloxetine HCl in Women of Different Demographic Characteristics and Co-Morbidities With Stress Urinary Incontinence: Evaluation of Efficacy and Safety
Brief Title: Safety and Effectiveness Study of Duloxetine HCl in Women of Different Backgrounds With Stress Urinary Incontinence Who May Also Have Other Various Medical Conditions.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8363; F1J-US-SBCD
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-07-25 (Estimated); Status verified 2006-07

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine HCl

SUMMARY:
The purpose of the trial is to study the safety and effectiveness of duloxetine HCl in women of different backgrounds with stress urinary incontinence who may also have other various medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years or older who have for the 3 months prior to study entry at least 1 episode per week of stress urinary incontinence or stress predominant urinary incontinence defined as twice as many stress as urge urinary incontinence episodes per week.
* Women of non-childbearing potential by reason of hysterectomy, surgical or natural menopause. Women of childbearing potential should be using a medically accepted means of contraception.
* Must provide informed consent.
* Must not have urinary tract infection at screening.

Exclusion Criteria:

* Sensitivity to duloxetine
* Unstable medical conditions
* Pregnancy
* Acute liver damage
* Suicidal in the opinion of the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000
Dates: Start 2004-02; Study Completion 2005-07

PRIMARY OUTCOMES:
Percent change in weekly incontinence episode frequency as noted by patient diaries from baseline to endpoint in Hispanic women and also in African American women with SUI or stress predominant mixed urinary incontinence

SECONDARY OUTCOMES:
Baseline to endpoint analysis for the Patient Global Impression of Improvement, Incontinence Quality of Life, and pad use as noted by patient diaries

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Indianapolis, Indiana, United States